CLINICAL TRIAL: NCT03721510
Title: A Phase 1/2a Open Label Study of the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of PGT121, VRC07-523LS and PGDM1400 Monoclonal Antibodies in HIV-uninfected and HIV-infected Adults
Brief Title: A Phase 1/2a Study of PGT121, VRC07-523LS and PGDM1400 Monoclonal Antibodies in HIV-uninfected and HIV-infected Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Orlando Immunology Center (Other); Houston AIDS Research Team (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IAVI T003
Record Dates: First submitted 2018-03-16; First posted 2018-10-26 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: HIV/AIDS
Keywords: HIV; AIDS; Monoclonal antibodies; Neutralizing antibodies; Analytical treatment interruption
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1A (Active Comparator): HIV-uninfected volunteers receiving one IV infusion
  Interventions: Biological: PGT121 + VRC07-523LS
- Group 1B (Active Comparator): HIV-uninfected volunteers receiving one IV infusion
  Interventions: Biological: PGT121 + VRC07-523LS + PGDM1400
- Group 2 (Active Comparator): HIV-infected volunteers on ART receiving three or six IV infusions
  Interventions: Biological: PGT121 + VRC07-523LS + PGDM1400

INTERVENTIONS:
Biological: PGT121 + VRC07-523LS — PGT121 + VRC07-523LS, dose 30 mg/kg each, given intravenously
  Arms: Group 1A
Biological: PGT121 + VRC07-523LS + PGDM1400 — PGT121 + VRC07-523LS + PGDM1400, dose 20 mg/kg each, given intravenously
  Arms: Group 1B; Group 2

SUMMARY:
This is a Phase 1/2a open label study to evaluate the safety, tolerability, pharmacokinetics and anti-viral activity of PGT121, VRC07-523LS and PGDM1400 for HIV prevention and therapy.

DETAILED DESCRIPTION:
This is a Phase 1/2a open label study to evaluate the safety, tolerability, pharmacokinetics and anti-viral efficacy of PGT121, VRC07-523LS and PGDM1400 antibodies for HIV prevention and therapy. PGT121, VRC07-523LS and PGDM1400 are recombinant human IgG1 monoclonal antibodies that target a V3 glycan-dependent epitope region of the HIV envelope protein and the CD4 binding site (CD4bs) of the HIV envelope protein. PGT121, VRC07-523LS and PGDM1400 mAbs were chosen for this study because of their potency, their ability to neutralize a wide array of cross-clade HIV viruses in a complementary pattern, and their proven antiviral activity in animal studies, e.g., their capacity to robustly prevent and treat simian-human immunodeficiency virus (SHIV) in rhesus monkeys.

The potency and breadth of PGT121, VRC07-523LS and PGDM1400 raise the possibility that monoclonal antibodies may be effective for HIV prophylaxis at low doses and against global viruses. Neutralization sensitivity profiles are complementary; and the combination of these mAbs with unique epitope specificities will provide experience assessing the potential additive, synergistic, or antagonistic properties of two bNAbs given sequentially.

ELIGIBILITY:
1. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
2. In the opinion of the Principal Investigator or designee and based on Assessment of Informed Consent Understanding results, has understood the information provided and potential impact and/or risks linked to IV infusion and participation in the trial; written informed consent will be obtained from the volunteer before any study-related procedures are performed.
3. All volunteers born female engaging in sexual activity that could lead to pregnancy must commit to use an effective method of contraception from the day of the first IV infusion of investigational product until 6 months following the final investigational product administration
4. All sexually active volunteers born male, regardless of reproductive potential, must be willing to consistently use an effective method of contraception from the day of investigational product administration until at least 6 months following the final investigational product administration to avoid exposure of partners to investigational product in ejaculate, and to prevent conception with female partners.
5. All volunteers born female must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Procedures and must test negative prior to investigational product administration.
6. All volunteers born female must agree not to donate eggs (ova, oocytes) for the purpose of assisted reproduction until 6 months after the final investigational product administration. Volunteers born male must agree not to donate sperm until 6 months after final investigational product administration.
7. Willing to forgo donations of blood and/or any other tissues, including bone marrow, during the study and, for those HIV-uninfected volunteers who test HIV-positive due to investigational product administration, until the anti-HIV antibody titers become undetectable.

Specific inclusion criteria for HIV-uninfected volunteers (Group 1):

1. Healthy male or female, including transgender, volunteers, as assessed by a medical history, physical exam, and laboratory test
2. At least 18 years of age on the day of screening and has not reached his or her 51st birthday on the day of signing the Informed Consent Document
3. Willing to undergo HIV testing, risk reduction counseling and receive HIV test results
4. Low risk for HIV infection for 12 months prior to study participation and willing to maintain low-risk behavior for the duration of the trial

Specific inclusion criteria for HIV-infected volunteers (Group 2):

1. At least 18 years of age on the day of screening and has not reached his or her 66th birthday on the day of signing the Informed Consent Document
2. Confirmed HIV-1 infection (HIV Ab+ or HIV RNA+) by documentation in the medical records or in-clinic HIV testing
3. CD4 ≥ 400 cells/µl
4. On antiretroviral therapy for a minimum of 24 months, with plasma HIV-1 RNA levels of < 50 copies/ml for at least 12 months as documented in the medical records, and with a viral load < 50 copies / ml at time of screening (within 56 days prior to IP administration). ART must not have been initiated during the acute phase of the infection as suggested by the available medical history and laboratory data from the time of the diagnosis. Note: ART is defined as a regimen including > 2 compounds, e.g., 2x nucleoside reverse transcriptase inhibitors plus either non-nucleoside reverse transcriptase inhibitor or protease inhibitor or integrase inhibitor.
5. If on an NNRTI-based regimen, willing to switch to an integrase inhibitor containing regimen for 4 weeks prior to discontinuing ART
6. No history of AIDS-defining illness within the past 5 years
7. No history of CD4 nadir <200 cells/ul
8. Under care of an HIV healthcare provider 5.6 Exclusion Criteria

Exclusion criteria for all volunteers:

1. Any clinically significant acute or chronic medical condition, other than HIV infection, that is considered progressive or in the opinion of the investigator makes the volunteer unsuitable for participation in the study.
2. Any clinically relevant abnormality on history or examination including history of immunodeficiency (other then HIV infection) or autoimmune disease; use of systemic corticosteroids, immunosuppressive, anticancer, or other medications considered significant by the investigator within the previous 6 months. The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least 6 weeks prior to enrollment in this study.
3. If born female, pregnant, lactating or planning a pregnancy during the period of screening through completion of the study.
4. In the past 6 months a history of alcohol or substance use, including marijuana, judged by the Investigator to potentially interfere with volunteer study compliance.
5. Bleeding disorder that was diagnosed by a physician. Note: A volunteer who states that he or she has easy bruising or bleeding, but does not have a formal diagnosis and has intramuscular injections and blood draws without any adverse experience, is eligible.
6. History of a splenectomy.
7. Receipt of live attenuated vaccine within the previous 30 days or planned receipt within 30 days after administration of investigational product; or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after infusion with investigational product (exception is live attenuated influenza vaccine within 14 days).
8. Receipt of blood transfusion or blood-derived products within the previous 3 months.
9. Participation in another clinical trial of an investigational product currently, within the previous 3 months or expected participation during this study. Note: receipt of placebo in a clinical trial in the previous 3 months will not exclude a volunteer from participation if documentation is available and the Medical Monitor gives approval.
10. Prior receipt of an investigational HIV vaccine candidate, monoclonal antibody or polyclonal immunoglobulin. Note: receipt of placebo in a previous HIV vaccine or monoclonal antibody trial will not exclude a volunteer from participation if documentation is available and the Medical Monitor gives approval.
11. History of severe local or systemic reactogenicity to injections or IV infusion (e.g., anaphylaxis, respiratory difficulties, angioedema).
12. Psychiatric condition that compromises safety of the volunteer and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
13. If, in the opinion of the Principal Investigator, it is not in the best interest of the volunteer to participate in the trial.
14. Seizure disorder: a volunteer who has had a seizure in the last 3 years is excluded.
15. Body mass index ≥ 35 or ≤ 18.5.
16. Infectious disease: chronic hepatitis B infection (HbsAg), current hepatitis C infection (HCV Ab positive and HCV RNA positive) or interferon-alfa treatment for chronic hepatitis C infection in the past year, chlamydia, gonorrhea, or active syphilis.
17. A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
18. Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic, antiviral or antifungal therapy within 30 days prior to enrollment.
19. Any of the following abnormal laboratory parameters listed below:

Hematology

* Hemoglobin < 10.5 g/dL in females; hemoglobin <11.0 g/dL in males
* Absolute Neutrophil Count (ANC): ≤ 1000/mm3
* Platelets: < 100,000 mm3 or ≥ 550,000/mm3 Chemistry
* AST ≥ 1.5 x ULN
* ALT ≥ 1.5 x ULN
* Total bilirubin ≥ 1.1 x ULN
* Alkaline phosphatase ≥ 1.5 x ULN
* Albumin ≤ 3.0 g/dL (equivalent to ≤ 30 g/L)
* Estimated Glomerular filtration rate (GFR) < 60 ml/min according to the Cockcroft Gault formula for creatinine clearance

  * Male: (140 - age in years) x (wt in kg) = CLcr (ml/min) / 72 x (serum creatinine in mg/dL)
  * Female: (140 - age in years) x (wt in kg) x 0.85 = CLcr (mL/min) / 72 x (serum creatinine in mg/dL)

Urinalysis: Any of the following abnormal findings if consistent with clinically significant disease:

* Protein = 2+ or more
* Blood = 2+ or more (not due to menses)

Specific exclusion criteria for HIV-uninfected volunteers (Group 1):

1. Confirmed HIV-1 infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability - Proportion of volunteers with moderate or greater reactogenicity | 3 days post infusion for each infusion
  Proportion of volunteers with moderate or greater reactogenicity (i.e., solicited adverse events) for 3 days following each IV infusion of PGT121, VRC07-523LS and PGDM1400 as assessed using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, July 2017, or the Common Terminology Criteria for Adverse Events (CTCAE,) Version 5.0 27 November 2017 (for reactogenicity observed within the first 24 hours post-infusion.)
Safety and Tolerability - Proportion of volunteers with adverse events (AEs) | 56 days
  Proportion of volunteers with adverse events (AEs), including safety laboratory (biochemical, hematological) parameters, during the 56 days following IV infusion of PGT121, VRC07-523LS and PGDM1400 that are moderate or greater, and/or considered related to PGT121 and/or VRC07-523LS and/or PGDM1400 as assessed using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, or the Common Terminology Criteria for Adverse Events (CTCAE,) Version 5.0 27 November 2017 (for reactogenicity observed within the first 24 hours post-infusion.)
Safety and Tolerability - Proportion of volunteers with serious adverse events (SAEs) | Up to 44 weeks
  Proportion of volunteers with serious adverse events (SAEs) throughout the study period following IV infusion(s) of PGT121, VRC07-523LS and PGDM1400 that are considered related to PGT121 and/or VRC07-523LS and/or PGDM1400 as assessed using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, or the Common Terminology Criteria for Adverse Events (CTCAE,) Version 5.0 27 November 2017 (for reactogenicity observed within the first 24 hours post-infusion.)
Pharmacokinetics - Elimination half-life (t1/2) | Up to 44 weeks
  Pharmacokinetics following IV infusion of PGT121, VRC07-523LS and PGDM1400 in HIV-uninfected and HIV-infected adults:
  • Elimination half-life (t1/2)
Pharmacokinetics - Clearance (CL/F) | Up to 44 weeks
  Pharmacokinetics following IV infusion of PGT121, VRC07-523LS and PGDM1400 in HIV-uninfected and HIV-infected adults:
  • Clearance (CL/F)
Pharmacokinetics - Volume of distribution (Vz/F) | Up to 44 weeks
  Pharmacokinetics following IV infusion of PGT121, VRC07-523LS and PGDM1400 in HIV-uninfected and HIV-infected adults:
  • Volume of distribution (Vz/F)
Pharmacokinetics - Area under the concentration decay curve (AUC) | Up to 44 weeks
  Pharmacokinetics following IV infusion of PGT121, VRC07-523LS and PGDM1400 in HIV-uninfected and HIV-infected adults:
  • Area under the concentration decay curve (AUC)

SECONDARY OUTCOMES:
Antiviral Activity - Proportion of volunteers who meet ART re-initiation criteria | Up to 44 weeks
  Proportion of volunteers who meet ART re-initiation criteria (defined as plasma HIV-1 RNA ≥ 1000 copies/ml and/or CD4 count < 300 cells/μl) on two consecutive measurements following ART interruption in Group 2
Antiviral Activity - Time to meeting ART re-initiation criteria | Up to 44 weeks
  Time to meeting ART re-initiation criteria (plasma HIV-1 RNA level ≥ 1000 copies/ml, CD4+ T cell count < 300 cells/ μl in two consecutive measurements) following ART interruption in Group 2
mAb serum levels at the time of viral rebound in Group 2 | Up to 44 weeks
  Serum levels of PGT121 at time of viral rebound
mAb serum levels at the time of viral rebound in Group 2 | Up to 44 weeks
  Serum levels of VRC07-523LS at time of viral rebound
mAb serum levels at the time of viral rebound in Group 2 | Up to 44 weeks
  Serum levels of PGDM1400 at time of viral rebound
CD4+ T cell count | Up to 44 weeks
  Change in CD4+ T cell count and frequency compared to baseline as measured by single platform flow cytometry in HIV-infected adults following IV infusion of PGT121, VRC07-523LS and PGDM1400.
Effects of PGT121, VRC07-523LS and PGDM1400 on viral escape mutations in rebound viruses | Up to 44 weeks
  Phylogenetic comparison of viruses grown from PBMCs collected from volunteers while on ART to rebound viruses collected after ART interruption (Group 2)
Anti-PGT121 antibodies | Up to 44 weeks
  Serum anti-PGT121 antibody titers
Anti-VRC07-523LS antibodies | Up to 44 weeks
  Serum anti-VRC07-523LS antibody titers
Anti-PGDM1400 antibodies | Up to 44 weeks
  Serum anti-PGDM1400 antibody titers

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orlando Immunology Center, Orlando, Florida
  - Center for Virology and Vaccine Research/ Clinical Trials Unit/ BIDMC, Boston, Massachusetts
  - Houston AIDS Research Team (HART), Houston, Texas

REFERENCES:
- [Derived] Julg B, Walker-Sperling VEK, Wagh K, Aid M, Stephenson KE, Zash R, Liu J, Nkolola JP, Hoyt A, Castro M, Serebryannyy L, Yanosick K, Speidel T, Borducchi EN, Murzda T, Maxfield L, Arduino R, McDermott AB, Gama L, Giorgi EE, Koup RA, Seaman MS, Rolle CP, DeJesus E, Li W, Korber B, Barouch DH. Safety and antiviral effect of a triple combination of HIV-1 broadly neutralizing antibodies: a phase 1/2a trial. Nat Med. 2024 Dec;30(12):3534-3543. doi: 10.1038/s41591-024-03247-5. Epub 2024 Sep 12. PMID 39266747
- See also: Related Info — http://iavi.org